CLINICAL TRIAL: NCT02220894
Title: A Randomized, Open Label, Phase III Study of Overall Survival Comparing Pembrolizumab (MK-3475) Versus Platinum Based Chemotherapy in Treatment Naïve Subjects With PD-L1 Positive Advanced or Metastatic Non-Small Cell Lung Cancer (Keynote 042)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Platinum-Based Chemotherapy for Participants With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Advanced or Metastatic Non-Small Cell Lung Cancer (MK-3475-042/KEYNOTE-042)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-042; 152877 (Registry Identifier: JAPIC-CTI); MK-3475-042 (Other: Merck Protocol Number); KEYNOTE-042 (Other: Merck); 2014-001473-14 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PD-1; PD1; PD-L1; PDL1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments.
  Interventions: Biological: pembrolizumab
- SOC Treatment (Active Comparator): Participants receive carboplatin target dose Area Under Curve (AUC) 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + paclitaxel 200 mg/m^2 IV on Day 1 of every 21-day cycle (Q3W) for a maximum of 6 cycles OR carboplatin target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + pemetrexed 500 mg/m^2 IV on Day 1 Q3W for a maximum of 6 cycles; participants with non-squamous histologies may go on to receive optional treatment with pemetrexed 500 mg/m^2 IV on Day 1 Q3W.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pemetrexed

INTERVENTIONS:
Biological: pembrolizumab
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: carboplatin
  Other Names: PARAPLATIN®
  Arms: SOC Treatment
Drug: paclitaxel
  Other Names: TAXOL®
  Arms: SOC Treatment
Drug: pemetrexed
  Other Names: ALIMTA®
  Arms: SOC Treatment

SUMMARY:
In this study, participants with programmed cell death ligand 1 (PD-L1)-positive non-small cell lung cancer (NSCLC) will be randomized to receive single agent pembrolizumab for up to 35 treatments or standard of care (SOC) platinum-based chemotherapy (carboplatin + paclitaxel or carboplatin + pemetrexed for 4 to 6 21-day cycles). Participants in the platinum-based chemotherapy arms with non-squamous tumor histologies may receive pemetrexed maintenance therapy after the 4 to 6 cycles of chemotherapy. The primary study hypothesis is that pembrolizumab prolongs overall survival (OS) compared to SOC chemotherapy.

DETAILED DESCRIPTION:
Pembrolizumab-treated participants, who attain a confirmed complete response (CR) or who stop trial treatment after 35 administrations of study medication for reasons other than disease progression or intolerability, may consider stopping trial treatment. These participants may be eligible for re-treatment with pembrolizumab monotherapy after they have experienced radiographic disease according to protocol-defined criteria. Response or progression in the Second Course Phase will not count towards the objective response rate (ORR) and progression free survival (PFS) endpoints in this trial.

The global study for MK-3475-042 enrolled 1274 participants. Of the 1274 total participants enrolled in the global study, 92 were also enrolled in the China extension study for MK-3475-042 (NCT03850444).

ELIGIBILITY:
Inclusion criteria:

* Histologically- or cytologically-confirmed diagnosis of advanced or metastatic NSCLC
* PD-L1 positive tumor
* Measureable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Life expectancy of at least 3 months
* No prior systemic chemotherapy for the treatment of the participant's advanced or metastatic disease (treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 6 months prior to diagnosis of advanced or metastatic disease)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function
* No prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy
* Submission of formalin-fixed diagnostic tumor tissue (in the case of participants having received adjuvant systemic therapy, the tissue should be taken after completion of this therapy)
* Female participants of childbearing potential must have a negative urine or serum pregnancy test and must be willing to use two adequate barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapeutic agents used in the study
* Male participants with a female partner(s) of child-bearing potential must be willing to use two adequate barrier methods of contraception from screening through 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapeutic agents used in the study

Exclusion criteria:

* Epidermal growth factor receptor (EGFR)-sensitizing mutation and/or is echinoderm microtubule-associated protein-like 4(EML4) gene/anaplastic lymphoma kinase (ALK) gene fusion positive
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study therapy
* No tumor specimen evaluable for PD-L1 expression by the central study laboratory
* Squamous histology and received carboplatin in combination with paclitaxel in the adjuvant setting
* Is receiving systemic steroid therapy ≤3 days prior to the first dose of study therapy or receiving any other form of immunosuppressive medication with the exception of daily steroid replacement therapy
* The NSCLC can be treated with curative intent with either surgical resection and/or chemoradiation
* Expected to require any other form of systemic or localized antineoplastic therapy while on study
* Any prior systemic cytotoxic chemotherapy, biological therapy or major surgery within 3 weeks of the first dose of study therapy; received lung radiation therapy >30 Gy within 6 months of the first dose of study therapy
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Known central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Had allogeneic tissue/solid organ transplantation
* Interstitial lung disease or history of pneumonitis that has required oral or IV steroids
* Has received or will receive a live vaccine within 30 days prior to the first study therapy (seasonal flu vaccines that do not contain live vaccine are permitted)
* Active infection requiring intravenous systemic therapy
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1274 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] de Castro G Jr, Kudaba I, Wu YL, Lopes G, Kowalski DM, Turna HZ, Caglevic C, Zhang L, Karaszewska B, Laktionov KK, Srimuninnimit V, Bondarenko I, Kubota K, Mukherjee R, Lin J, Souza F, Mok TSK, Cho BC. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy as First-Line Therapy in Patients With Non-Small-Cell Lung Cancer and Programmed Death Ligand-1 Tumor Proportion Score >/= 1% in the KEYNOTE-042 Study. J Clin Oncol. 2023 Apr 10;41(11):1986-1991. doi: 10.1200/JCO.21.02885. Epub 2022 Oct 28. PMID 36306479
- [Derived] Halmos B, Burke T, Kalyvas C, Insinga R, Vandormael K, Frederickson A, Piperdi B. Indirect comparison of pembrolizumab monotherapy versus nivolumab + ipilimumab in first-line metastatic lung cancer. Immunotherapy. 2022 Apr;14(5):295-307. doi: 10.2217/imt-2021-0273. Epub 2022 Jan 25. PMID 35073727
- [Derived] Wu YL, Zhang L, Fan Y, Zhou J, Zhang L, Zhou Q, Li W, Hu C, Chen G, Zhang X, Zhou C, Dang T, Sadowski S, Kush DA, Zhou Y, Li B, Mok T. Randomized clinical trial of pembrolizumab vs chemotherapy for previously untreated Chinese patients with PD-L1-positive locally advanced or metastatic non-small-cell lung cancer: KEYNOTE-042 China Study. Int J Cancer. 2021 May 1;148(9):2313-2320. doi: 10.1002/ijc.33399. Epub 2020 Dec 9. PMID 33231285
- [Derived] Weng X, Luo S, Lin S, Zhong L, Li M, Xin R, Huang P, Xu X. Cost-Utility Analysis of Pembrolizumab Versus Chemotherapy as First-Line Treatment for Metastatic Non-Small Cell Lung Cancer With Different PD-L1 Expression Levels. Oncol Res. 2020 Mar 27;28(2):117-125. doi: 10.3727/096504019X15707883083132. Epub 2019 Oct 14. PMID 31610828
- [Derived] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1275 participants randomized (pembrolizumab=638, chemotherapy=637), 1 participant assigned to receive pembrolizumab died prior to randomization and was randomized in error. The intent to treat population was defined as participants alive at the time of randomization, so the actual randomized population included 637 participants in each arm.
Pre-assignment Details: Pembrolizumab-treated participants, who attained a confirmed complete response (CR) or who stopped trial treatment after 35 administrations of study medication for reasons other than disease progression or intolerability, could consider stopping trial treatment. These participants may have been eligible for re-treatment with pembrolizumab monotherapy after they had experienced radiographic disease as per protocol-defined criteria.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 every 3 weeks (Q3W) for a maximum of 35 cycles (21-day cycles). Some participants may have been eligible for re-treatment with pembrolizumab monotherapy after they had experienced radiographic disease as per protocol-defined criteria.
- Chemotherapy (Standard of Care [SOC] Treatment): Participants received carboplatin at target dose Area Under Curve (AUC) 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + paclitaxel 200 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles) OR carboplatin target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles). Participants with non-squamous histologies received optional additional maintenance treatment with pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W
Period: Overall Study
Arm/Group | Pembrolizumab | Chemotherapy (Standard of Care [SOC] Treatment)
Started | 637 (1 additional participant was randomized in error) | 637
Treated | 636 | 615
Completed | 0 | 0
Not Completed | 637 | 637
Not completed — Adverse Event | 127 | 74
Not completed — Death | 418 | 508
Not completed — Lost to Follow-up | 0 | 4
Not completed — Site Terminated by Sponsor | 2 | 0
Not completed — Participation in Study Terminated by Sponsor | 80 | 41
Not completed — Withdrawal by Parent/Guardian | 0 | 1
Not completed — Withdrawal by Subject | 10 | 9

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants who were alive at the time of randomization and had a Tumor Proportion Score (TPS) ≥1%.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by IV infusion on Day 1 Q3W for a maximum of 35 cycles (21-day cycles)
- Chemotherapy (SOC Treatment): Participants received carboplatin at target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + paclitaxel 200 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles) OR carboplatin target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles). Participants with non-squamous histologies received optional additional maintenance treatment with pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment) | Total
Number analyzed (Participants) | 637 | 637 | 1274
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (9.9) | 63.1 (9.4) | 62.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 185 | 372
  Male | 450 | 452 | 902
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 5 | 15
  Asian | 189 | 187 | 376
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 13 | 23
  White | 398 | 412 | 810
  More than one race | 30 | 19 | 49
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair or Grade 5: Dead.
  Participants
    ECOG PS=0 | 197 | 192 | 389
    ECOG PS=1 | 439 | 445 | 884
    ECOG PS=2 | 1 | 0 | 1
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a tumor proportion score (TPS) were classified as follows: ≥50% = PD-L1 strongly positive; 1-49% = PD-L1 weakly positive; and <1% = PD-L1 negative.
  Participants
    TPS=≥50% | 299 | 300 | 599
    TPS=20-49% | 114 | 105 | 219
    TPS=1-19% | 224 | 232 | 456
    TPS=<1% | 0 | 0 | 0
Tumor Histology [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous. The tumor histology determined potential treatment regimen.
  Participants
    Squamous | 242 | 249 | 491
    Non-squamous | 395 | 388 | 783

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: OS was determined for participants with a TPS of ≥50% and was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was OS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The OS for participants with a TPS ≥50% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 299 | 300
Months | 20.0 [15.9 to 24.2] | 12.2 [10.4 to 14.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0003, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.58 to 0.86] — Hazard ratio based on Cox regression model with treatment as a covariate stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1), and histology (squamous vs. non-squamous)

2. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: OS was determined for participants with a TPS of ≥20% and was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was OS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The OS for participants with a TPS ≥20% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 413 | 405
Months | 18.0 [15.4 to 21.9] | 13.0 [11.6 to 15.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0012, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.65 to 0.91] — Hazard ratio based on Cox regression model with treatment as a covariate stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1), PD-L1 expression status (TPS=≥50% vs. TPS=1-49%) and histology (squamous vs. non-squamous)

3. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: OS was determined for participants with a TPS of ≥1% and was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was OS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The OS for participants with a TPS ≥1% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 637 | 637
Months | 16.4 [14.0 to 19.7] | 12.1 [11.3 to 13.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0013, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.71 to 0.93] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: PFS was determined for participants with a TPS of ≥50% and was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was PFS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The PFS for participants with a TPS ≥50% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 299 | 300
Months | 6.5 [5.9 to 8.5] | 6.4 [6.2 to 7.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0260, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 1.00] — Hazard ratio based on Cox regression model with treatment as a covariate stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1) and histology (squamous vs. non-squamous)

5. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: PFS was determined for participants with a TPS of ≥20% and was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was PFS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The PFS for participants with a TPS ≥20% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 413 | 405
Months | 6.2 [5.1 to 7.4] | 6.7 [6.3 to 8.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.2134, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.80 to 1.10] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: PFS was determined for participants with a TPS of ≥1% and was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was PFS in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The PFS for participants with a TPS ≥1% is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 637 | 637
Months | 5.4 [4.3 to 6.2] | 6.6 [6.3 to 7.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.7964, Log Rank — One-sided p-value based on stratified log-rank test; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.93 to 1.19] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: ORR was determined for participants with a TPS of ≥50%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was ORR in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The percentage of participants who had a TPS ≥50% and who experienced a CR or PR is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 299 | 300
Percentage of participants | 39.1 [33.6 to 44.9] | 32.0 [26.8 to 37.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0353, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in percentages=0 vs. H1: difference in percentages >0; Difference in Percentage (DP) = 7.0, 95% CI 2-sided [-0.6 to 14.6] — DP for pembrolizumab vs. chemotherapy based on Miettinen & Nurminen method stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1) and histology (squamous vs. nonsquamous)

8. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: ORR was determined for participants with a TPS of ≥20%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was ORR in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The percentage of participants who had a TPS ≥20% and who experienced a CR or PR is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 413 | 405
Percentage of participants | 33.2 [28.6 to 37.9] | 28.9 [24.5 to 33.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.0744, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in percentages=0 vs. H1: difference in percentages >0; Difference in Percentage (DP) = 4.6, 95% CI 2-sided [-1.7 to 10.9] — DP for pembrolizumab vs. chemotherapy based on Miettinen & Nurminen method stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1), PD-L1 expression status (TPS=≥50% vs. TPS=1-49%) and histology (squamous vs. non-squamous)

9. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: ORR was determined for participants with a TPS of ≥1%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The efficacy hypothesis was analyzed using a sequential testing strategy that involved testing a hypothesis only if the superiority of pembrolizumab over chemotherapy was established for all the preceding hypotheses. The order of testing was ORR in participants with TPS≥50%, then with TPS≥20%, and finally with TPS≥1%. The percentage of participants who had a TPS ≥1% and who experienced a CR or PR is presented.
Time Frame: Up to approximately 44 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 637 | 637
Percentage of participants | 27.2 [23.7 to 30.8] | 26.5 [23.1 to 30.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Superiority; p = 0.4060, Stratified Miettinen and Nurminen — One-sided p-value for testing. H0: difference in percentages=0 vs. H1: difference in percentages >0; Difference in Percentage (DP) = 0.6, 95% CI 2-sided [-4.2 to 5.4] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 38 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 636 | 615
Participants | 608 | 606

11. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 35 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 636 | 615
Participants | 126 | 93

ADVERSE EVENTS:
Time Frame: Up to approximately 93 months
Description: Population: All participants receiving ≥1 dose of study treatment. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab Second Course: Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment) | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 528/637 | 582/637 | 18/34
Serious Adverse Events (participants affected / at risk) | 261/636 | 193/615 | 8/34
Other Adverse Events (participants affected / at risk) | 535/636 | 577/615 | 21/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=636) | Chemotherapy (SOC Treatment) (N=615) | Pembrolizumab Second Course (N=34)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 16 (23) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 1 (1)
Death (General disorders) | 9 (9) | 5 (5) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 49 (54) | 34 (41) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (5) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 5 (7) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 16 (17) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Normochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 4 (4) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 8 (8) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pleural infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood prolactin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=636) | Chemotherapy (SOC Treatment) (N=615) | Pembrolizumab Second Course (N=34)
Anaemia (Blood and lymphatic system disorders) | 102 (124) | 253 (332) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 10 (17) | 35 (63) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (9) | 85 (177) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 59 (86) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 37 (38) | 4 (4) | 1 (1)
Hypothyroidism (Endocrine disorders) | 76 (99) | 10 (10) | 3 (5)
Constipation (Gastrointestinal disorders) | 78 (98) | 131 (168) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 74 (94) | 78 (107) | 3 (5)
Nausea (Gastrointestinal disorders) | 73 (98) | 195 (407) | 1 (1)
Vomiting (Gastrointestinal disorders) | 50 (62) | 106 (167) | 0 (0)
Asthenia (General disorders) | 69 (92) | 81 (110) | 2 (3)
Chest pain (General disorders) | 56 (61) | 43 (52) | 1 (1)
Fatigue (General disorders) | 101 (129) | 129 (193) | 0 (0)
Malaise (General disorders) | 15 (15) | 32 (49) | 1 (1)
Pyrexia (General disorders) | 64 (82) | 52 (63) | 1 (1)
Pneumonia (Infections and infestations) | 39 (40) | 30 (35) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 46 (62) | 32 (41) | 1 (1)
Alanine aminotransferase increased (Investigations) | 66 (89) | 72 (97) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 62 (83) | 57 (87) | 3 (3)
Neutrophil count decreased (Investigations) | 6 (6) | 89 (239) | 0 (0)
Platelet count decreased (Investigations) | 7 (7) | 65 (144) | 0 (0)
Weight decreased (Investigations) | 67 (71) | 48 (49) | 4 (4)
White blood cell count decreased (Investigations) | 5 (7) | 77 (228) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 108 (127) | 134 (209) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (26) | 32 (43) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 (109) | 87 (162) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 61 (70) | 43 (51) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (37) | 70 (135) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (36) | 34 (40) | 0 (0)
Dizziness (Nervous system disorders) | 25 (28) | 39 (49) | 0 (0)
Insomnia (Psychiatric disorders) | 34 (38) | 45 (51) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 107 (128) | 66 (72) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 105 (120) | 72 (81) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 45 (62) | 23 (25) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 138 (139) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 67 (83) | 22 (23) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 72 (82) | 43 (52) | 1 (4)
Hypertension (Vascular disorders) | 41 (49) | 14 (17) | 1 (1)
Nasopharyngitis (Infections and infestations) | 26 (37) | 21 (26) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 16 (18) | 33 (40) | 0 (0)
Oedema peripheral (General disorders) | 32 (33) | 36 (50) | 1 (1)
Bronchitis (Infections and infestations) | 30 (34) | 23 (25) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 39 (46) | 30 (35) | 2 (2)
Headache (Nervous system disorders) | 44 (58) | 51 (62) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 5 (6) | 52 (62) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 43 (55) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT02220894/Prot_SAP_001.pdf